CLINICAL TRIAL: NCT02692508
Title: Morphological and Functional Changes and Prognosis of Subjects With Unexplainable Precordial Deep T-wave Inversion Without Apical Wall Thickness> 15mm
Brief Title: Prognosis of Subjects With Unexplainable Precordial Deep T-wave Inversion Without Wall Thickness> 15mm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other); Peking Union Medical College Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Minjie Lu, Vice Director of Magnetic Resonance Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: AHCM001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cardiomyopathy; Hypertrophic
Keywords: cardiovascular MRI; apical hypertrophic cardiomyopathy; giant negative T-wave; wall thickness; Nuclear Magnetic Resonance; Early Diagnosis; Prognosis
MeSH Terms: conditions — Cardiomyopathies; Hypertrophy; Apical Hypertrophic Cardiomyopathy; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators sought to evaluate the morphological and functional changes and prognosis of participants with unexplainable precordial deep T-wave inversion on ECG and with apical thickness less than 15mm. The conduction of this study was largely due to the increased clinical requirement, which reflected the increased awareness among physicians of missed AHCM.

DETAILED DESCRIPTION:
Apical hypertrophic cardiomyopathy (AHCM) is a special form of non obstructive hypertrophic cardiomyopathy (HCM), in which the hypertrophy of myocardium predominantly involves the apex of the left ventricle (LV). Generally, patients with AHCM show obvious negative T waves on precordial leads on electrocardiogram (ECG). However, clinically some patients present dramatic T-wave inversion with the apical thickness less than the diagnostic criteria of AHCM. In order to get a moderate diagnosis, these participants may undergo lengthy investigation with implications for lifestyle modifications and increase the health care expenses. The investigators wonder they may share their fate with patients who have overt AHCM. Further study of these patients is needed for a proper diagnosis and treatment.

In conventional diagnostic criteria published by American heart association (AHA)/American college of cardiology foundation (ACCF) in 2011, or European society of cardiology (ESC) in 2014, the LV wall thickness≥15 mm is the unified diagnostic criteria of HCM. These guidelines, however, did not give additional regulations or instructions for the diagnosis of AHCM. It is suspected that these criteria may be too strict for AHCM, as the normal left ventricular wall thins towards the apex and the normal values are lower naturally in the apical versus the basal segments.

Comparing with echocardiography, the superior spatial and temporal resolution of CMR makes it more sensitive to diagnose AHCM at earlier stage, much earlier than the appearance of "ace-of-spades" configuration. In a previous study, only 60% of patients with apical segmental hypertrophy that were confirmed by CMR were diagnosed by echocardiography. Echocardiography has its technical limitations for assessing apex due to the limited regional spatial resolution. Additionally, CMR can offer prognostic features, such as apical scar and apical aneurysms.

The investigators thus sought to evaluate the morphorage and functional changes and prognosis of participants with unexplainable precordial deep T-wave inversion on ECG and with apical thickness less than 15mm.The conduction of this study was largely due to the increased clinical requirement, which reflected the increased awareness among physicians of missed AHCM.

ELIGIBILITY:
Inclusion Criteria:

* Standard 12-lead electrocardiography showing deep T-wave inversion, most prominent in the anterolateral leads (V3-V5 leads) with the negative T wave voltage ≥5mm.
* Without evidence of coronary artery disease, or diameter stenosis ≥50% in one or more coronary vessels.
* Asymmetrical LV hypertrophy confined to the LV apex below the papillary muscle level; end-diastolic apical wall thickness <15mm with the apical to basal posterior wall thickness ratio <1.5.

Exclusion Criteria:

* Subjects who were not in sinus rhythm;
* Patients with T-wave inversion in ≤ 2 contiguous leads, concomitant bundle branch block or QRS>80 ms or QTC>440 ms were excluded.
* Blood pressure ≥140/90mmHg.
* Severe valvular lesion, pericardial disease, cardiac tumor, immunological or metabolic disease involving heart.
* History of cardiac surgery.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: subjects with unexplainable precordial deep T-wave inversion on ECG and with apical thickness less than 15mm
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
apical hypertrophic cardiomyopathy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Lu, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Failure Society of America; Heart Rhythm Society; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 13;124(24):2761-96. doi: 10.1161/CIR.0b013e318223e230. Epub 2011 Nov 8. No abstract available. PMID 22068435
- [Result] Gersh BJ, Maron BJ, Bonow RO, Dearani JA, Fifer MA, Link MS, Naidu SS, Nishimura RA, Ommen SR, Rakowski H, Seidman CE, Towbin JA, Udelson JE, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American Society of Echocardiography; American Society of Nuclear Cardiology; Heart Failure Society of America; Heart Rhythm Society; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons. 2011 ACCF/AHA guideline for the diagnosis and treatment of hypertrophic cardiomyopathy: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 13;124(24):e783-831. doi: 10.1161/CIR.0b013e318223e2bd. Epub 2011 Nov 8. No abstract available. PMID 22068434
- [Result] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Result] Dawson DK, Maceira AM, Raj VJ, Graham C, Pennell DJ, Kilner PJ. Regional thicknesses and thickening of compacted and trabeculated myocardial layers of the normal left ventricle studied by cardiovascular magnetic resonance. Circ Cardiovasc Imaging. 2011 Mar;4(2):139-46. doi: 10.1161/CIRCIMAGING.110.960229. Epub 2010 Dec 30. PMID 21193690
- [Result] Lee PT, Dweck MR, Prasher S, Shah A, Humphries SE, Pennell DJ, Montgomery HE, Payne JR. Left ventricular wall thickness and the presence of asymmetric hypertrophy in healthy young army recruits: data from the LARGE heart study. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):262-7. doi: 10.1161/CIRCIMAGING.112.979294. Epub 2013 Jan 10. PMID 23307776
- [Result] Lu M, Zhao S, Jiang S, Yin G, Wang C, Zhang Y, Liu Q, Cheng H, Ma N, Zhao T, Chen X, Huang J, Zou Y, Song L, He Z, An J, Renate J, Xue H, Shah S. Fat deposition in dilated cardiomyopathy assessed by CMR. JACC Cardiovasc Imaging. 2013 Aug;6(8):889-98. doi: 10.1016/j.jcmg.2013.04.010. Epub 2013 Jul 10. PMID 23850250
- [Result] Lu M, Zhao S, Yin G, Jiang S, Zhao T, Chen X, Tian L, Zhang Y, Wei Y, Liu Q, He Z, Xue H, An J, Shah S. T1 mapping for detection of left ventricular myocardial fibrosis in hypertrophic cardiomyopathy: a preliminary study. Eur J Radiol. 2013 May;82(5):e225-31. doi: 10.1016/j.ejrad.2012.12.014. Epub 2013 Jan 17. PMID 23333530
- [Result] Florian A, Masci PG, De Buck S, Aquaro GD, Claus P, Todiere G, Van Cleemput J, Lombardi M, Bogaert J. Geometric assessment of asymmetric septal hypertrophic cardiomyopathy by CMR. JACC Cardiovasc Imaging. 2012 Jul;5(7):702-11. doi: 10.1016/j.jcmg.2012.03.011. PMID 22789938